CLINICAL TRIAL: NCT05472246
Title: The Effect of Virtual Reality Headset on Anxiety, Sedation Need and Patient Satisfaction in Oncological Patients Scheduled for Port Catheter Implantation
Brief Title: The Effect of Virtual Reality Headset on Anxiety, Sedation Need
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mesut Aslan (Other)
Responsible Party: Sponsor-Investigator, Mesut Aslan, Asistant Doctor, Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital
Organization: Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VRsedation
Record Dates: First submitted 2022-07-19; First posted 2022-07-25 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Anxiety Postoperative; Anesthesia; Patient Satisfaction
Keywords: VR; Anxiety; PortCatheter
MeSH Terms: conditions — Patient Satisfaction; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Our study is a prospective, randomized, controlled, single-center study involving 200 patients aged 18-70 years who are scheduled for port catheter implantation procedure in Dr Siyami Ersek Thoracic Heart and Vascular Surgery Training and Research Hospital Thoracic Surgery Clinic. The patients will be randomly divided into 2 groups and one group will be shown relaxing videos (nature scenes) by wearing a VR headset in addition to the routine anesthesia procedure, while the control group will undergo the routine anesthesia procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental): VR group will be shown relaxing videos (nature scenes) by wearing a VR headset in addition to the routine anesthesia procedure.
  Interventions: Device: Wearing a virtual reality headset
- Control group (No Intervention): Control group will undergo the routine anesthesia procedure.

INTERVENTIONS:
Device: Wearing a virtual reality headset — VR group will be shown relaxing videos (nature scenes) by wearing a VR headset in addition to the routine anesthesia procedure
  Arms: VR group

SUMMARY:
In our clinic, our aim is to evaluate the effects of virtual reality technology on pain, anxiety, and additional anesthesia needs in patients undergoing port catheter implantation.

DETAILED DESCRIPTION:
The patients will be randomly divided into 2 groups and one group will be shown relaxing videos (nature scenes) by wearing a VR headset in addition to the routine anesthesia procedure, while the control group will undergo the routine anesthesia procedure.

All patients are taken to the operating room, patients will be informed about the study and VR headsets, informed consent forms will be obtained, and preoperative anxiety levels will be evaluated with the STAI (state-transit anxiety inventory) questionnaire. Patients will be monitored in accordance with American Society of Anesthesiologist (ASA) standards within the routine anesthesia practices and vital signs (ECG: Electrocardiogram, Non-invasive SAP: Systolic arterial pressure, DAP: Diastolic arterial pressure, MAP: mean arterial pressure, HR: heart rate, SpO2: peripheral oxygen saturation) will be monitored and an intravenous cannula will be placed. In the VR group, the patient will wear the VR headset right before the surgical procedure starts and will be removed after the last surgical suture is performed. If the patient initially consents but wishes to remove the VR headset during the procedure or if the anesthesiologist considers it necessary, the headsets can be removed, and these patients will be recorded. An anesthesiologist and a study member will be present in the operating room to adjust VR headsets and help with technical issues. The anesthesiologist will apply routine anesthesia protocols to both groups, administer any additional medications deemed necessary, and any additional medications will be recorded. Each patient will receive midazolam 0.05 mg/kg IV and fentanyl 1 mcg/kg IV immediately after intravenous cannula placement as part of the routine sedation protocol of anesthesia. The sedation level of the patients will be targeted at 2-3 levels according to the Ramsey Sedation Scale and 1-2.5 mg/kg/hr IV propofol infusion will be given. The surgical team will administer local anesthesia. The onset of anesthesia will be recorded when midazolam is administered, the completion will be recorded when the patient awakens, and the duration of anesthesia will be recorded as the time between these two events. The beginning of surgery, the moment the surgeon performs the local anesthesia, the end of the surgery, the end of the last suture and the duration of the surgery will be recorded as the time between these two events. The postoperative anxiety level will be assessed with the STAI (State-Trait Anxiety Inventory) questionnaire 1 hour after the end of surgery (T2) in the post-anesthesia care unit (PACU). In this study, no additional monitoring and drug administration will be performed, except for the procedures included in the routine sedation protocol of anesthesia.

Primary data are the need for additional anesthetics (total intraoperative propofol dose in mg, additional opiod dose in mcg) and anxiety levels. Secondary data are hemodynamic data (MAP, HR, SpO2 will be recorded every 10 minutes), patient satisfaction, time to put on and adjust VR headsets, number of patients who refuse VR headsets, number of patients who remove VR headsets before the procedure ends. Demographic data (age, gender, weight, height, body mass index-BMI), ASA and comorbidities, duration of surgery and anesthesia will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Oncological Patients
2. Patients aged 18-70 years scheduled for port catheter implantation
3. ASA 1-3 patients

Exclusion Criteria:

1. Patients under 18 years of age and over 70 years of age.
2. Patients with open wounds or infections around the face and eyes.
3. Patients diagnosed with epilepsy or with a history of seizures for any reason.
4. Patients using a pacemaker or an implanted medical device.
5. Patients who do not speak Turkish.
6. Patients with a history of psychiatric and neurological disorders.
7. Patients with a history of vertigo.
8. Patients who are allergic to any of the drugs to be used in the study.
9. Patients who have taken sedatives in the last 24 hours.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
additional anesthetics | peroperative
  the need for additional anesthetics (total intraoperative propofol dose in mg, additional opiod dose in mcg)
anxiety levels change | 15 minutes before operatian and after 1 hour of operation
  After all patients are taken to the operating room, patients will be informed about the study and VR headsets, informed consent forms will be obtained, and anxiety levels will be evaluated with the STAI (state-transit anxiety inventory) questionnaire. The postoperative anxiety level will be assessed with the STAI (State-Trait Anxiety Inventory) questionnaire 1 hour after the end of surgery (T2) in the post-anesthesia care unit (PACU).

SECONDARY OUTCOMES:
blood pressure change | Peroperative
  Mean arterial blood pressure:mm Hg will be recorded every 10 minutes
heart rate change | Peroperative
  heart rate: beat/minute will be recorded every 10 minutes
SpO2 change | Peroperative
  SpO2:%0-100 will be recorded every 10 minutes
patient satisfaction | after 1 hour of operation
  Patient satisfaction will be assessed and recorded using a 5-point patient satisfaction scale. (1: Extremely dissatisfied, 2: Dissatisfied, 3: Unknown or Uncertain, 4: Satisfied, 5: Extremely satisfied)
time to put on and adjust VR headsets | Preoperative
  minute
number of patients who refuse VR headsets | preoperative
  number
number of patients who remove VR headsets before the procedure ends | Peroperative
  number
duration of surgery and anesthesia | Peroperative
  minute

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Yavuzel, Principal Investigator — Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital; Tülin Satılmış, Principal Investigator — Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital; Mesut Aslan, Principal Investigator — Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital
Locations (1):
- Dr.Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)